CLINICAL TRIAL: NCT03899766
Title: Animal Assisted Activity, Clowns and Music for the Reduction of Distress and Pain in Children During Venipuncture
Brief Title: Support Activities for the Reduction of Distress and Pain in Children During Venipuncture
Status: Completed | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Laura Vagnoli, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: SupportActivities_Venipuncture
Record Dates: First submitted 2018-12-24; First posted 2019-04-02 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Venipuncture
Keywords: pain, procedural; child; anxiety
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Animal Assisted Intervention: children interact and play with the expert of Animal Assisted Intervention (AAI) and his/her trained dog in the waiting room and then, are accompanied by a parent (as standard care) and the AAI in the venipuncture room during and immediately after the procedure
  Interventions: Other: Animal Assisted Intervention
- Clowns: children interact and play with hospital clowns in the waiting room and then, are accompanied by a parent (as standard care) and the clown in the venipuncture room during and immediately after the procedure
  Interventions: Other: Clowns
- Musicians: children interact and play with a musician in the waiting room and then, are accompanied by a parent (as standard care) and the musician in the venipuncture room during and immediately after the procedure
  Interventions: Other: Musicians
- Non-clinical Conversation: children are accompanied by a parent in the waiting room and then in the venipuncture room during the procedure, thus receiving standard care

INTERVENTIONS:
Other: Animal Assisted Intervention — Operators of AAI and their dog meet the child and his/her parent in the waiting room and facilitates interaction using their professional characteristics. The interaction continue in the venipuncture room during the procedure and at its conclusion; in fact, the operators accompany the child and his/her parent outside the venipuncture room, to not abruptly interrupt the interaction.
  Groups: Animal Assisted Intervention
Other: Clowns — Hospital clowns meet the child and his/her parent in the waiting room and facilitates interaction using their professional characteristics. The interaction continue in the venipuncture room during the procedure and at its conclusion; in fact, the operators accompany the child and his/her parent outside the venipuncture room, to not abruptly interrupt the interaction.
  Groups: Clowns
Other: Musicians — Musicians meet the child and his/her parent in the waiting room and facilitates interaction using their professional characteristics. The interaction continue in the venipuncture room during the procedure and at its conclusion; in fact, the operators accompany the child and his/her parent outside the venipuncture room, to not abruptly interrupt the interaction.
  Groups: Musicians

SUMMARY:
To evaluate the efficacy of Health Support Activities (Animal Assisted Intervention, Clows, Musicians) in the reduction of pain and distress in children undergoing venipuncture.

Hypothesis: the investigators expect a reduction in in pain and distress.

DETAILED DESCRIPTION:
Venipuncture is one of the most unpleasant procedures for children. Previous studies demonstrated the effectiveness of distraction techniques in reducing anxiety and pain but no one compares the specific activities of animals assisted intervention (AAI), clowns and musicians for this procedure.

In the Hospital involved in the present study, venipuncture service has a week schedule for Health Support Activities. In specific days children can benefit of Health Support Activities as part of routine care.

Aims of the present study are: evaluate efficacy of AAI, clowns and musicians in the reduction of childrens' distress and pain during venipuncture with respect of a control group undergoing venipuncture in the days where Health Support Activities are not scheduled; compare distress and pain levels between groups; evaluate caregiver's anxiety and its influence on child pain and distress; explore parents' and staff opinion.

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* scheduled to venipuncture
* Italian speaking

Exclusion Criteria:

* cognitive and/or developmental impairment

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Outpatiens reffering to hospital for venipuncture
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Distress | Distress assessment is one for every participant and begins when child enter in the venipuncture room and lasts until the child exit the venipuncture room, in the day of recruitment. .
  Brief Behavioral Distress Scale - BBDS is an observational measure that assess children's procedure-related distress with 12 discrete component steps involved in venipuncture, in order to observe specific demands for compliance on the child during the procedure. Observers record the occurrence or nonoccurrence of the target behaviors during each step. Operational definitions of the target behaviors for each category are: 1) Non interfering Distress Behaviors; 2) Potentially Interfering Distress Behaviors; 3) Interfering Distress Behaviors. The number of steps in which a behavior occur is summed and divided by the total number of steps, then multiplied by 100 to yield percentage of steps with occurrence scores for each behavioral category. The number of steps in which behaviors from any of the three distress behavior categories occur is summed and divided by the total number of steps multiplied by three, then multiplied by 100 to obtain the Total Distress Score.
Pain perception 3-6 years old | Pain assessment is one for every participant, measured immediately after the child exit the venipuncture room, in the day of recruitment
  Numerical scales, based on age, Wong Baker Scale. The Wong Baker Faces Pain Rating Scale (Wong & Baker, 1998) is a self-report scale for children older than 3 years old, that shows a sequence of faces ranging from a happy face at 0 level, that means "No hurt", to a crying face at 10th level, that means "Hurts worst".
Pain perception from 7 years old | Pain assessment is one for every participant, measured immediately after the child exit the venipuncture room, in the day of recruitment
  Numerical scale, Visual Analogue Scale - VAS. VAS is used from the age of 7 years old, is a self-report numerical scale ranging from 0, that means "No pain", to 10, that means "worst pain".

SECONDARY OUTCOMES:
Parent's state and trait anxiety | Parent's anxiety assessment is one for every participant, measured in the waiting room before child enters in the venipuncture room, in the day of recruitment
  Self-report scale (State-Trait Anxiety Inventory - STAI). The STAI is a self-report anxiety behavioral instrument for adults. It consists of two separate subscales: one assessing trait anxiety (baseline, Y1), the other assessing the state anxiety (situational, Y2). Each subscale is composed by 20 items, rated on a 4-points Likert scale and separately analyzed. Total score for each subscale range from 20 to 80, with higher scores denoting higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Messeri, MD, Study Director — Meyer Children's Hospital IRCCS; Laura Vagnoli, MSc, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (1):
- Meyer Children's Hospital, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Decision has to be shared with the Clinical Trial Office of the Hospital

REFERENCES:
- [Background] Bijttebier P, Vertommen H. The Impact of Previous Experience on Children's Reactions to Venepunctures. J Health Psychol. 1998 Jan;3(1):39-46. doi: 10.1177/135910539800300103. PMID 22021341
- [Background] Caprilli S, Anastasi F, Grotto RP, Scollo Abeti M, Messeri A. Interactive music as a treatment for pain and stress in children during venipuncture: a randomized prospective study. J Dev Behav Pediatr. 2007 Oct;28(5):399-403. doi: 10.1097/DBP.0b013e31811ff8a7. PMID 18049324
- [Background] Duff AJ. Incorporating psychological approaches into routine paediatric venepuncture. Arch Dis Child. 2003 Oct;88(10):931-7. doi: 10.1136/adc.88.10.931. PMID 14500318
- [Background] Goodenough B, Thomas W, Champion GD, Perrott D, Taplin JE, von Baeyer CL, Ziegler JB. Unravelling age effects and sex differences in needle pain: ratings of sensory intensity and unpleasantness of venipuncture pain by children and their parents. Pain. 1999 Mar;80(1-2):179-90. doi: 10.1016/s0304-3959(98)00201-2. PMID 10204730
- [Background] Kaminsky M. (2002). Play and Pets: The Physical and Emotional Impact of Child-Life and Pet Theraphy on Hospitalized Children. Children's Health Care, 31(4), 321-335.
- [Background] Kennedy RM, Luhmann J, Zempsky WT. Clinical implications of unmanaged needle-insertion pain and distress in children. Pediatrics. 2008 Nov;122 Suppl 3:S130-3. doi: 10.1542/peds.2008-1055e. PMID 18978006
- [Background] Kolk AM, van Hoof R, Fiedeldij Dop MJ. Preparing children for venepuncture. The effect of an integrated intervention on distress before and during venepuncture. Child Care Health Dev. 2000 May;26(3):251-60. doi: 10.1046/j.1365-2214.2000.00145.x. PMID 10921442
- [Background] Meiri N, Ankri A, Hamad-Saied M, Konopnicki M, Pillar G. The effect of medical clowning on reducing pain, crying, and anxiety in children aged 2-10 years old undergoing venous blood drawing--a randomized controlled study. Eur J Pediatr. 2016 Mar;175(3):373-9. doi: 10.1007/s00431-015-2652-z. Epub 2015 Oct 16. PMID 26475347
- [Background] Treurnicht Naylor K, Kingsnorth S, Lamont A, McKeever P, Macarthur C. The effectiveness of music in pediatric healthcare: a systematic review of randomized controlled trials. Evid Based Complement Alternat Med. 2011;2011:464759. doi: 10.1155/2011/464759. Epub 2010 Sep 30. PMID 20976017
- [Background] Tsao JC, Lu Q, Myers CD, Kim SC, Turk N, Zeltzer LK. Parent and child anxiety sensitivity: relationship to children's experimental pain responsivity. J Pain. 2006 May;7(5):319-26. doi: 10.1016/j.jpain.2005.12.004. PMID 16632321
- [Background] Uman LS, Birnie KA, Noel M, Parker JA, Chambers CT, McGrath PJ, Kisely SR. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2013 Oct 10;(10):CD005179. doi: 10.1002/14651858.CD005179.pub3. PMID 24108531
- [Background] Uman LS, Chambers CT, McGrath PJ, Kisely S. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD005179. doi: 10.1002/14651858.CD005179.pub2. PMID 17054243
- [Background] Birnie KA, Noel M, Chambers CT, Uman LS, Parker JA. Psychological interventions for needle-related procedural pain and distress in children and adolescents. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005179. doi: 10.1002/14651858.CD005179.pub4. PMID 30284240
- [Background] Vagnoli L, Caprilli S, Vernucci C, Zagni S, Mugnai F, Messeri A. Can presence of a dog reduce pain and distress in children during venipuncture? Pain Manag Nurs. 2015 Apr;16(2):89-95. doi: 10.1016/j.pmn.2014.04.004. Epub 2014 Nov 4. PMID 25439114
- [Background] Wolyniez I, Rimon A, Scolnik D, Gruber A, Tavor O, Haviv E, Glatstein M. The effect of a medical clown on pain during intravenous access in the pediatric emergency department: a randomized prospective pilot study. Clin Pediatr (Phila). 2013 Dec;52(12):1168-72. doi: 10.1177/0009922813502257. Epub 2013 Sep 11. PMID 24028842
- [Background] Yoo H, Kim S, Hur HK, Kim HS. The effects of an animation distraction intervention on pain response of preschool children during venipuncture. Appl Nurs Res. 2011 May;24(2):94-100. doi: 10.1016/j.apnr.2009.03.005. Epub 2009 Jul 15. PMID 20974061